CLINICAL TRIAL: NCT06639633
Title: Investigation of the Effect of Magnified Carpal Bones Produced With High Resolution 3D Resin Printer on Students' Theoretical and Practical Anatomy Grades and Learning Levels
Brief Title: 3D Printed Enlarged Carpal Models for Anatomy Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assist. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-FTR-RK-09
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Anatomical Pathological Condition; Educational Problems
Keywords: Resin; Segmentation
MeSH Terms: conditions — Pathological Conditions, Anatomical

STUDY DESIGN:
Intervention Model Description: Prospective parallel group with single-blinded design
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3D Printed Model Group Enlarged %100 (Other): carpal bone models printed on a 3D resin printer and enlarged by 100% will be used for students' anatomy practical training. Each student will examine the models with direct manipulation for 15 minutes after the theoretical lecture.
  Interventions: Other: Anatomy Training with Enlarged %100 3D Printed Carpal Model Group
- 3D Printed Model Group Enlarged %50 (Other): carpal bone models printed on a 3D resin printer and enlarged by 50% will be used for students' anatomy practical training. Each student will examine the models with direct manipulation for 15 minutes after the theoretical lecture.
  Interventions: Other: Anatomy Training with Enlarged %50 3D Printed Carpal Model Group
- Control Group (Active Comparator): Standard carpal bone models will be used for student's anatomical practical training. Each student will examine the models with direct manipulation for 15 minutes after the theoretical lecture.
  Interventions: Other: Anatomy Training with Conventional Carpal Models

INTERVENTIONS:
Other: Anatomy Training with Enlarged %100 3D Printed Carpal Model Group — After completing the general terminology part of the anatomy education in the first year, the participants will be recruited without moving on to the hand section of the upper extremity. Participants will undergo a 2-hour extra-curricular training, 60 minutes theoretical and 60 minutes practical. The training period will consist of 60 minutes of practical and theoretical lectures to be the same as the time allocated in the normal curriculum of the region. A 60-minute theoretical lecture on the anatomy of the carpal bone supported by 2-dimensional anatomical pictures will be given to both groups at the same time. Then they will take the practical lesson with carpal bones printed with 100% magnification on a 3D printer for 60 minutes.
  Arms: 3D Printed Model Group Enlarged %100
Other: Anatomy Training with Enlarged %50 3D Printed Carpal Model Group — After completing the general terminology part of the anatomy education in the first year, the participants will be recruited without moving on to the hand section of the upper extremity. Participants will undergo a 2-hour extra-curricular training, 60 minutes theoretical and 30 minutes practical. The training period will consist of 60 minutes of practical and theoretical lectures to be the same as the time allocated in the normal curriculum of the region. A 60-minute theoretical lecture on the anatomy of the carpal bone supported by 2-dimensional anatomical pictures will be given to both groups at the same time. Then they will take the practical lesson with carpal bones printed with 50% magnification on a 3D printer for 60 minutes.
  Arms: 3D Printed Model Group Enlarged %50
Other: Anatomy Training with Conventional Carpal Models — After completing the general terminology part of the anatomy education in the first year, the participants will be recruited without moving on to the hand section of the upper extremity. Participants will undergo a 2-hour extra-curricular training, 60 minutes theoretical and 60 minutes practical. The training period will consist of 60 minutes of practical and theoretical lectures to be the same as the time allocated in the normal curriculum of the region. A 60-minute theoretical lecture on the anatomy of the carpal bone supported by 2-dimensional anatomical pictures will be given to both groups at the same time. They will then have a 60 minutes practical lesson with a standard sized printed model.
  Arms: Control Group

SUMMARY:
3D modeling enables medical professionals or students to better understand complex structures. In many studies, 3D printed models have been used in the training, treatment and surgery of medical disciplines such as neuroscience, cardiovascular surgery and otolaryngology. In addition, 3D modeling allows patients' magnetic resonance imaging (MRI) and computed tomography (CT) images to be transferred to 3D printers to print these complex structures.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Titmus stereopsis score >40 arc/s

Exclusion Criteria:

* Previous experience of carpal bones models either in real world or virtual reality
* History of upper extremity trauma in past 6 months
* Total or partial eye sight lost

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Quiz Scores | 1 hour
  In order to measure the anatomical terminology and general knowledge of the students, a general test will be applied before the pre-test and the groups will be distributed according to this test score. Then, a total of 20 theoretical and 20 practical questions of 10 questions each will be prepared to be used in the pre-test and post-test. The questions will be under the headings of bony prominences, neighborhood, important structures, adhesion sites and function.

SECONDARY OUTCOMES:
Model rating with Visual Analogue Scale | 1 hour
  After the completion of the final exam, a visual analog scale will be used to evaluate the model. Participants will mark the level of detail, appropriateness of weight, ease of learning, ease of grasping and direct manipulation, and ease of distinguishing details/details on a 10 cm long straight line.
Academic motivation Scale | 1 hour
  The Test-Taking Motivation questionnaire scale will be used to assess the motivation of the participants. The scale consists of 22 questions and 7 subscales and assesses amotivation, intrinsic and extrinsic motivation.
Test Anxiety Inventory | 1 hour
  A short version of the 5-item Test Anxiety Inventory consisting of 5 questions will be used to examine whether there is a change in the amount of anxiety students experience during the exam.
Enjoyment and Ease of Use Assessmen | 1 hour
  Participants will fill out a feedback questionnaire regarding the learning instruments using visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Kurul, Ph.D, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
data of this study will be available after the publication of the study and will be usable upon citing the related article
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the publication of the study
Access Criteria: upon citing the related article